CLINICAL TRIAL: NCT04898491
Title: Validity and Reliability Study of the Pain Indicator Behavior Scale Adapted to Measure Pain in Critically Ill Patients With Acquired Brain Damage, Non-communicative and With an Artificial Airway (ESCID-DC).
Brief Title: Validity and Reliability Study of the Pain Indicator Behavior Scale-Brain Damage (ESCID-DC)
Acronym: ESCID-DC
Status: Recruiting | Type: Observational
Sponsor: Candelas Lopez Lopez (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Candelas Lopez Lopez, RN, MSc, PhD, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Other Study IDs: ESCID-DC
Record Dates: First submitted 2021-05-11; First posted 2021-05-24 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Pain; Brain Injuries; Behavior
Keywords: Pain; Brain injury; Brain damage; Intensive Critical Unit; Nursing
MeSH Terms: conditions — Pain; Brain Injuries; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Pain assessment using a behavioral scale — The pain of the subjects will be evaluated by two independent observers and with a blind result between them, coinciding with the application of two painful procedures used in routine practice: suction of tracheal secretions and the pressure in the nail bed by means of a pressure algometer. In addition, a painless procedure will also be performed to establish an element of control with the procedures painful. This will consist of the application of gentle friction with a cloth gauze, on a part of healthy skin tissue of the patient. The measurement will be performed twice for each patient and procedure depending on the level of sedation, so that the first measurement will be performed with a deeper sedation level and the second with a change in sedation level to moderate-mild.
  In turn, the pain assessment will be carried out in three moments: first or baseline measurement, during the application of the painless and 15 minutes after finishing the procedures.

SUMMARY:
A multicentre observational study to validate the adaptation of the Pain Indicator Behavior Scale (ESCID) for patients with acquired Brain Damage (ESCID-DC), as a measuring instrument.

DETAILED DESCRIPTION:
Non-commercial study. The study complies with the ethical principles of the Declaration of Helsinki, the recommendations of Good Clinical Practice (GCP) and current legislation.

The study has been approved with a favorable opinion by the CEIm of the Hospital Universitario 12 de Octubre.

Written consent will be requested from the participants and / or their relatives / representatives to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age equal to or greater than 18 years.
2. Inability to communicate verbally or motor.
3. Have a artificial airway.
4. Informed consent of the family member or representative of the patient.

Exclusion Criteria:

1. Previous pathology of cognitive impairment.
2. Previous brain injury.
3. Previous psychiatric disorder.
4. Previous dementia.
5. Previous chronic substance abuse.
6. Previous chronic diabetics.
7. Previous spinal cord injury.
8. Previous severe polyneuropathy (diagnosed or suspected).
9. Confirmed diagnosis of brain death.
10. Continuous infusion of muscle relaxants and / or barbiturate coma.
11. Level of deep sedation (RASS -5).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acquired brain damage (ACD) admitted to the Intensive Critical Care (ICU) of the aforementioned hospitals, who comply with all the inclusion criteria and none of the exclusion criteria for the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
To assess the construct validity and the reliability | 30 months
  Number of patients with Brain Damage, non-communicative and artificial airway that manifest pain behaviors included in the Pain Indicator Behavior Scale-Brain Damage

SECONDARY OUTCOMES:
To assess pain from different procedures with ESCID-DC scale | 30 months
  Pain score of patients before, during and after performing two procedures documented as painful (aspiration of tracheal secretions and application of pressure to the nail bed), common in the routine care of critically ill patients, and a procedure not painful (gentle friction with a cloth gauze on skin tissue) using the Indicator Behavior Scale of Pain in a Patient with Brain Damage (ESCID-DC)
To assess pain from different procedures with NCS-R scale | 30 months
  Pain score of patients before, during and after performing two procedures documented as painful (aspiration of tracheal secretions and application of pressure to the nail bed), common in the routine care of critically ill patients, and a procedure not painful (gentle friction with a cloth gauze on skin tissue) using the Nociception Coma Scale-Revised (NCS-R)
To analyze the scale under different etiology of brain damage | 30 months
  Pain score of patients with different etiology of brain damage (ischemic, traumatic and / or post-anoxic encephalopathy)
To analyze the scale under different levels of consciousness | 30 months
  Pain score of patients with different levels of consciousness (severe: Glasgow Coma Score <9 / moderate: Glasgow Coma Score 9-13 / mild: Glasgow Coma Score 14-15)
To analyze the scale under different degrees of sedation | 30 months
  Pain score of patients with different degrees of sedation (deep sedation: Richmond Agitation-Sedation Scale (RASS) Score -5, -4 / moderate sedation: Richmond Agitation-Sedation Scale (RASS) Score -3 and/or light sedation Richmond Agitation-Sedation Scale (RASS) Score -2, -1)

CONTACTS AND LOCATIONS:
Overall Officials: Candelas López-López, PhD, Study Chair — Emergency and Trauma Intensive Care Unit. Hospital Universitario 12 de Octubre
Locations (1):
- Emergency and Trauma Intensive Care Unit. Hospital Universitario 12 de Octubre, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez-Lopez C, Latorre-Marco I, Sanchez-Sanchez MDM, Sarabia-Cobo CM, Solis-Munoz M, Perez-Perez T, Roldan-Merino J, Robleda-Font G. Content Validation of the Behavioural Indicators of Pain Scale in Critically Ill Patients With Acquired Brain Injury: A Delphi Study. Nurs Crit Care. 2025 May;30(3):e70053. doi: 10.1111/nicc.70053. PMID 40417781
- [Derived] Lopez-Lopez C, Latorre-Marco I, Perez-Perez T, Sarabia-Cobo CM, Solis-Munoz M, Sanchez-Sanchez MDM, Arranz-Esteban A, Frade-Mera MJ, Temprano-Vazquez S, Robleda-Font G. Validity and Reliability of the Behavioural Indicators of Pain Scale Adapted to Patients With Acquired Brain Injury: ESCID-DC Study Protocol. J Adv Nurs. 2025 Aug;81(8):5143-5150. doi: 10.1111/jan.16983. Epub 2025 Apr 18. PMID 40249752